CLINICAL TRIAL: NCT04546243
Title: A Retrospective Study Investigating Survival for High-grade Osteosarcoma Patients Who Had Achieved First Complete Surgical Remission (SCR) During Combined-modality Therapy in Two Hospitals Affiliated to Peking University
Brief Title: Osteosarcoma With Resectable Pulmonary Metastasis: A Retrospective Study
Status: Completed | Type: Observational
Sponsor: Peking University People's Hospital (Other)
Collaborators: Peking University Shougang Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: PKUPH-sarcoma 13
Record Dates: First submitted 2020-09-04; First posted 2020-09-11 (Actual); Last update posted 2020-12-04 (Actual); Status verified 2020-12

CONDITIONS: Osteosarcoma Metastatic; Pulmonary Disease; Resectable Sarcoma; Survival
Keywords: osteosarcoma; pulmonary metastasis; resectable; event-free survival
MeSH Terms: conditions — Lung Diseases; Osteosarcoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- osteosarcoma patients receiving resections
  Interventions: Procedure: resection group
- osteosarcoma patients receiving radiotherapy
  Interventions: Radiation: radiotherapy group

INTERVENTIONS:
Procedure: resection group — patients received VATS
  Groups: osteosarcoma patients receiving resections
Radiation: radiotherapy group — patients received radiotherapy
  Groups: osteosarcoma patients receiving radiotherapy

SUMMARY:
According to EURAMOS-1, 17% of osteosarcoma patients were considered to have metastases at diagnosis. In this selected cohort, the reported 5-year EFS from diagnosis of 28% compares well to previous results reported from unselected cohorts of patients with only lung metastases. Resection of pulmonary metastases from osteosarcoma is a treatment option which has been shown to correlate with survival benefit and cure in select individuals. These patients are best addressed in a multidisciplinary fashion, with the involvement of a thoracic surgeon with experience in pulmonary metastasectomy. At the same time, the goal of surgical resection of pulmonary metastases from osteosarcoma is to render the patient completely disease free. "Tumor debulking" or "cytoreductive surgery" with incomplete resection has not demonstrated any survival benefit for patients with pulmonary metastases. Thus open thoracotomy is more preferred than VATS. However over the last decade in China, thoracotomy has not been adopted generally. More patients had chosen VATS or even hypo-fractionation radiotherapy, such as gamma knife, cyber knife and so on as a local treatment method. This study aims to investigate the survival of consecutive patients who had achieved a first complete surgical remission (CR) during combined-modality therapy on neoadjuvant or adjuvant PKUPH-OS protocol so as to discuss reasonable local therapy for resectable pulmonary osteosarcoma metastatic lesions.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed high-grade osteosarcoma reviewed by the Pathology Committee of Peking University People's Hospital
* Pulmonary nodules by Chest CT confirmed by later scan as pulmonary metastasis
* A first complete remission (CR) had been achieved
* Intended first-line treatment included pre- and postoperative chemotherapy according to the PKUPH-OS protocol as well as local therapy of all operable lesions

Exclusion Criteria:

* Lost to follow up
* Patients with severe or uncontrolled medical disorders that could jeopardize the outcomes of the study. These confounding conditions included, cardiac clinical symptoms or disease with left ventricular ejection fraction<50%, and hypertension that could not be well controlled with antihypertensive drugs.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: This report includes all the patients with recurrences from a previously treated cohort of 678 consecutive, newly diagnosed patients with localized or primary metastatic high-grade osteosarcoma of the trunk or limbs registered onto the neoadjuvant studies of Peking University People's Hospital and Peking University Shougang Hospital between the end of 2009 and March 2020. Intended first-line treatment included pre- and postoperative chemotherapy according to the PKUPH-OS protocol , as well as surgery of all operable lesions. All protocols prescribed high-dose methotrexate, doxorubicin, cisplatin and ifosfamide in varying combinations.
Sampling Method: Non-Probability Sample
Enrollment: 127 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2020-10-01 (Actual); Study Completion 2020-11-01 (Actual)

PRIMARY OUTCOMES:
event-free survival | 2 year
  from local therapy of the pulmonary nodules to any events of progression of disease/last follow-up

SECONDARY OUTCOMES:
local recurrence rate | 2 year
  from local therapy of the pulmonary nodules to local recurrence/last follow-up
overall survival | 5 year
  from local therapy of the pulmonary nodules to death/last follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Wei Guo, M.D., Principal Investigator — Musculoskeletal Tumor Center of Peking University People's Hospital
Locations (2):
- China (2):
  - Peking University Shougang Hospital, Beijing, Beijing Municipality
  - Peking University People's Hospital, Beijing, Beijing Municipality

IPD SHARING:
Plan to Share IPD: No